CLINICAL TRIAL: NCT04930458
Title: Remineralization of Dentine Caries Using Nanosilver Fluoride and Casein Phosphopeptides-amorphous Calcium Phosphate (A Randomized Clinical Trial)
Brief Title: Remineralization of Dentine Caries Using Two Remineralizing Agents Which Are Nanosilver Fluoride and Casein phosphopeptides_amorphous Calcium Phosphate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, duaa jawad, Dentist.. master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dentine caries remineralizatio
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
Keywords: Dental caries remineralization; Nanosilver fluoride
MeSH Terms: conditions — Dental Caries | interventions — Sodium Fluoride; Bifluorid 12

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nanosilver fluoride group (Experimental): Nanosilver fluoride will be applied on carious lesion
  Interventions: Other: Nanosilver fluoride
- Sodium fluoride with casein phosphopeptides_Amorphous calcium phosphate group (Active Comparator): Sodium fluoride with casein phosphopeptides_Amorphous calcium phosphate will be applied on carios lesion
  Interventions: Other: Sodium fluoride with casein phosphopeptides amorphous calcium phosphate
- Sodium fluoride varnish group (Active Comparator): Sodium fluoride varnish will be applied on carios lesion
  Interventions: Other: Sodium fluoride varnish

INTERVENTIONS:
Other: Nanosilver fluoride — Nanosilver fluoride will be applied to the affected tooth in single application and then follow up after one and three months
  Arms: Nanosilver fluoride group
Other: Sodium fluoride with casein phosphopeptides amorphous calcium phosphate — Sodium fluoride with casein phosphopeptides amorphous calcium phosphatewill be applied to the affected tooth in single application and then follow up after one and three months
  Arms: Sodium fluoride with casein phosphopeptides_Amorphous calcium phosphate group
Other: Sodium fluoride varnish — Sodium fluoride varnish will be applied to the affected tooth in single application and then follow up after one and three months
  Arms: Sodium fluoride varnish group

SUMMARY:
The study is randomized controlled trial ...The null hypothesis suggests that there is no significant difference between nanosilver fluoride and sodium fluoride with Casein phosphopeptides_amorphous calcium phosphate in the remineralization of dental caries.

DETAILED DESCRIPTION:
the patients will be randomly assigned to one of three study groups the first group is nanosilver fluoride,the second is casein phosphopeptides_amorphous calcium phosphate and the third is sodium fluoride as positive control..the three material will be applied in single application with no repetition ..follow up after one and three month ..the patient should have at least one carious lesion(ICDASII code 5)

ELIGIBILITY:
* Clinical diagnosis of carious lesion
* participants should be free of any systemic diseases.

Exclusion Criteria:

* sensitivity to Silver or other heavy-metal ions or any milk-related allergies and medical conditions involving the kidneys.
* The tooth was excluded if it had pulp exposure, abscess/fistula, sensitivity to percussion

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of patient with arrested dental caries using international caries detection and assessment system II(ICDAS II) | Change in the state of dental caries after one and 3 months after topical application of nanosilver fluoride and sodium fluoride with casein phosphopeptides amorphous calcium phosphate
  The measure will be done using international caries detection and assessment system II (ICDAS II) criteria for diagnosing active and arrested caries by blunt probe.

CONTACTS AND LOCATIONS:
Overall Officials: Duaa Jawad, Principal Investigator — University of Baghdad
Locations (1):
- Alhur alriyahi specialized dental center, Karbala, Iraq